CLINICAL TRIAL: NCT05969457
Title: Effect of Preventive Analgesia by Injection of a Local Anesthetic Before Vaginal Incision for Hysterectomy by vNOTES Approach: Randomized, Double-blind Study
Brief Title: Effect of Preventive Analgesia by Injection of a Local Anesthetic Before Vaginal Incision for Hysterectomy by vNOTES Approach
Acronym: ANOTES
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHU de Rouen
Record Dates: First submitted 2023-07-17; First posted 2023-08-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Hysterotomy; Affecting Fetus
MeSH Terms: interventions — Ropivacaine; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experienced group (Experimental): Administration of Naropeine
  Interventions: Drug: Naropeine; Other: questionnaires
- Control group (Placebo Comparator): Administration of a saline solution
  Interventions: Other: questionnaires; Other: Placebo

INTERVENTIONS:
Drug: Naropeine — Local anesthesia with injection of Ropivacaine (20mL of ropivacaine 7.5 mg/mL, i.e. 150mg)
  Arms: Experienced group
Other: questionnaires — Numerical Rating scale Questionnaire FSFI Qustionnaire SF12 Questionnaire DN4
Other: Placebo — Injection of 20 mL of NaCl
  Arms: Control group

SUMMARY:
The research procedure is the injection of 20 mL of Ropivacaine solution (vs. saline) to create a paracervical block at the beginning of surgery, while the patient is already under general anesthesia.

This injection will take place 3 minutes before the vaginal incision, via 4 injection points. Injections are made 3 mm deep into the vaginal cul de sac.

Randomization takes place before surgery by vNOTES:

* Experienced group: Local anesthesia with injection of Ropivacaine (20mL of ropivacaine 7.5 mg/mL, i.e. 150mg) and general anesthesia
* Control group: Injection of 20mL of placebo (saline) and general anesthesia

In both groups, systematic intraoperative and postoperative analgesia will be identical.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 70 inclusive
* Patient scheduled for vNOTES surgery for total hysterectomy for benign pathology, whether or not associated with an adnexal procedure (unilateral or bilateral salpingectomy or adnexectomy (for cysts smaller than 6 cm)).
* Person having read and understood the information letter and signed the consent form
* Person affiliated to a social security scheme

Exclusion Criteria:

* Suspicion of malignant pathology
* History of rectal surgery
* History of pelvic inflammatory disease
* Suspicion of recto-vaginal endometriosis
* Virginity
* Contraindication to NAROPEINE 7.5 mg/mL, solution for injection in ampoule
* Contraindication to PROAMP SODIUM CHLORIDE 0.9%, solution for injection
* Patients on a low-salt diet
* History of more than 2 caesarean sections
* Estimated uterine size > 700 g according to the following formula y = 0.35x + 107 (x = a × b × c), based on measurements taken on preoperative imaging (MRI or ultrasound). a=longitudinal diameter, b=sagital diameter, c=transverse diameter.3
* BMI > 35
* Contraindication to analgesic molecules in intraoperative and postoperative protocols.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 108 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
pain after surgery | 4hours after surgery
  Pain will be assessed by the post-operative hospital nurse using a numerical rating scale (NRS) NRS score from 1 to 10 -> 10 correspoding to the worst pain

IPD SHARING:
Plan to Share IPD: No